CLINICAL TRIAL: NCT04883320
Title: Exploring the Role of Stem Cell Strategies for the Treatment of Chronic Asthma
Brief Title: Stem Cell Strategies for the Treatment of Chronic Asthma
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1175
Record Dates: First submitted 2021-04-30; First posted 2021-05-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Airway cells will be obtained from participants during bronchoscopy via biopsy, brush biopsy and bronchoalveolar lavage (BAL). To minimise discomfort the procedure will utilise the sedative midazolam and local anaesthetic lidocaine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- participants with no asthma: Have no evidence of any long term lung condition or any other disabling condition and they must not have had a chest infection in the preceding 4 weeks.
- participants with mild/moderate asthma
- participants with severe asthma

SUMMARY:
The study is a pilot/laboratory study comparing the effects of MSC conditioned media on samples of airway cells in 3 participant groups with mild/moderate asthma (5 participants), severe asthma (5 participants), or no asthma (5 participants).

DETAILED DESCRIPTION:
Asthma is a significant global health challenge with the prevalence of allergic asthma increasing by 1% each year. Atopic asthma is a complex disorder driven by cellular mechanisms in response to allergens. The response is two-fold; a chronic inflammatory response accompanied by remodelling of the respiratory airways. Airway remodelling is characterised by smooth muscle hypertrophy (and mucous gland) and hyperplasia, fibrosis of the sub-epithelium and reticular basement thickening, and epithelial damage. Over time the airway suffers remodelling due to thickening of the smooth muscle component which is in turn accompanied by irreversible fibrotic changes and a tendency towards treatment unresponsiveness. The inflammatory response on the other hand is characterised by IgE activation of mucous mast cells, infiltration of eosinophils, increased CD4+Th2 lymphocytes, and Type 2 cytokine secretion (e.g. IL13). The primary challenge in the development of new asthma treatments is to deliver long-lasting relief to the inflammatory response and also to 'repair' the remodelling associated with repeated asthmatic events. Mesenchymal stem cells (MSC), derived primarily from the bone marrow, have a multipotent differentiation potential (primarily bone, fat, and cartilage) and are currently in clinical trial for over 350 diseases and disorders. These include diverse areas such as ischemic stroke, graft vs. host disease, Crohns disease, and type 1 diabetes alongside anticipated applications related to the musculoskeletal system. Their application into the treatment of musculoskeletal damage relies primarily on functional incorporation (differentiation into the damaged tissue to repair in situ). In contrast their application in many other instances is due to their unique inherent characteristic, namely their immunomodulatory role. MSC secrete a wide range of growth factors and cytokines (the secretome) which have the capacity to silence immune reactions preventing T cell activation. In addition to this property the MSC secretome has also been shown to reverse the remodelling associated with fibrotic disease.

ELIGIBILITY:
Inclusion Criteria:

Men or women, age (18-70 years old), II. Lifelong never-smokers or ex-smokers (< 10 pack years). (1 pack year= 20 cigarettes/day for 1 year).

III. Must be competent to give written informed consent. IV. Female participants of child bearing potential must have a negative urine pregnancy test prior to bronchoscopy.

V Potential participants must meet the safety criteria to have a Spirometry test where necessary.

vi Must meet the safety criteria to have a bronchoscopy.

Asthmatic participants:

VI. Have a physician diagnosis of asthma. VII. All asthma patients will have either bronchodilator reversibility of ≥12% or 200 mL at screening, or historic data confirming bronchodilator reversibility or bronchial hyperreactivity to methacholine (PC20). Those without prior confirmed reversibility will have bronchodilator reversibility testing to salbutamol at screening and the asthma control questionnaire (ACQ) administered. Where reversibility to salbutamol is inconclusive a methacholine challenge will be performed.

VIII. Must have stable disease with no recent flare-ups (within 4 weeks). IX. Oxygen saturations whilst breathing room air must be > 90% (a measure of how well the lungs are providing oxygen to the body).

X. When blowing forcefully into a tube (forced expiratory volume or FEV), the patient must be able to blow out at least one litre of air in the first second (FEV1 > 1Litre).

Non-asthmatic participants:

XI. Have no physician diagnosis of asthma. XII. Have no evidence of any long term lung condition or any other disabling condition and they must not have had a chest infection in the preceding 4 weeks.

Exclusion Criteria:

I. Significant smoking history (>10 pack year). II. Significant lung co-morbidities III. Patient unable to give informed consent IV. History of myocardial infarction within the preceding 6 weeks V. Any subject with asthma who requires home oxygen will not be included for safety reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trial participants will be identified from those attending respiratory medicine outpatient clinics at the Royal Stoke University Hospital. Participants will donate samples of upper airway cells during bronchoscopy by biopsy, brush biopsy and bronchoalveolar lavage (BAL)
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-08-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The overall aim of this proposal is to determine the effects of adult stem cell products on asthmatic respiratory epithelium. | Through to study completion, average of one year
  Our primary objective is to determine this with in vitro models, where we will explore the utility of the MSC secretome in abrogating IgE and Type 2 cytokine driven immune responses and in reversing airway remodelling.

SECONDARY OUTCOMES:
Develop in virto models | Through to study completion, average of one year
  Our secondary objective is to develop in vitro models derived from patient materials obtained by brush and biopsied airway epithelium and bronchial airway cells via BAL from patients with established history of asthma and atopy and commercially sourced MSCs.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom